CLINICAL TRIAL: NCT03107052
Title: A Multicenter, Double-Blind, Double-Dummy Study to Explore the Long-Term Safety and Efficacy of TEV-48125 for the Prevention of Cluster Headache
Brief Title: A Study to Explore the Long-Term Safety and Efficacy of Fremanezumab (TEV-48125) for the Prevention of Cluster Headache
Acronym: ENFORCE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated after the episodic cluster study was terminated due to a pre specified futility analyses
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30058; 2016-003172-43 (EudraCT Number)
Record Dates: First submitted 2017-03-23; First posted 2017-04-11 (Actual); Results first posted 2020-05-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fremanezumab 225 mg Monthly (Experimental): Participants with ECH or CCH who received fremanezumab at 900 mg intravenous (IV) infusion at Week 0 and fremanezumab at 225 mg subcutaneous (SC) injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30056 or TV48125-CNS-30057, and participants with CCH who received fremanezumab at 675 mg SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30057; will receive fremanezumab at 225 mg SC injection monthly (approximately every 4 weeks, administered as single SC injection of fremanezumab at 225 mg [225 mg/1.5 milliliter {mL}] at Week 0 and 36; and 2 placebo SC injections at Weeks 0, 12, 24, and 36 for blinding in participants rolled over from Study TV48125-CNS-30056; fremanezumab at 225 mg as a single SC injection (225 mg/1.5 mL) at Week 0, 12, 24, and 36; 2 SC injections of placebo at Week 0 for blinding in participants rolled over from Study TV48125-CNS-30057) through Week 36 in this study.
  Interventions: Drug: Fremanezumab
- Fremanezumab 675/225 mg Monthly (Experimental): Participants with CCH who received placebo IV infusion and SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30057; will receive fremanezumab 675 mg SC injection as loading dose (administered as 3 SC injections of fremanezumab at 225 mg [225 mg/1.5 mL] at Week 0) followed by monthly (approximately every 4 weeks) fremanezumab at 225 mg SC injection (administered as single SC injection of fremanezumab at 225 mg [225 mg/1.5 mL] at Weeks 12, 24, and 36) through Week 36.
  Interventions: Drug: Fremanezumab
- Fremanezumab 675 mg Quarterly (Experimental): Participants with ECH who received fremanezumab at 675 mg SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study; or placebo IV infusion and SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30056; will receive fremanezumab at 675 mg SC injection quarterly (approximately every 12 weeks, administered as 3 SC injections of fremanezumab at 225 mg [225 mg/1.5 mL] at Weeks 0 an 36; and single placebo SC injections at Weeks 4, 8, 16, 20, 28, and 32 for blinding) through Week 36.
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab
  Other Names: TEV-48125

SUMMARY:
This is a 68-week study to evaluate the long-term safety and efficacy of fremanezumab in participants with cluster headache (CH). Participants who complete the pivotal studies TV48125-CNS-30056 (NCT02945046) and TV48125-CNS-30057 (NCT02964338) and enroll into the current study will visit the investigational center for investigational medicinal product (IMP) administration, safety and efficacy assessments, and blood and urine collections for pharmacokinetics, immunogenicity (anti-drug antibodies [ADAs]), and biomarker analyses. Participants will return to the investigational center for a follow-up visit to evaluate ADAs, fremanezumab concentrations, biomarkers, and safety (adverse events and concomitant medications) approximately 7.5 months after the last dose of IMP.

ELIGIBILITY:
Inclusion Criteria:

* The participant completes either the Phase 3 pivotal study for ECH (Study TV48125-CNS-30056) or the Phase 3 pivotal study for CCH (Study TV48125-CNS-30057) without important protocol deviations related to participant safety and participant compliance.
* Prior to 15 June 2018, participants from the ECH study and the CCH study were enrolled. After 15 June 2018, only participants who participated in the ECH study (Study TV48125-CNS-30056) will be enrolled for active treatment.
* In addition, participants who do not complete the pivotal efficacy studies, and participants who complete the pivotal efficacy studies but will not continue treatment during this long-term safety study, will be offered to enroll in this study for the purpose of evaluating ADAs, and safety (adverse events and concomitant medications) approximately 7.5 months after administration of the last dose of the IMP.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Any finding that, in the judgment of the investigator, is a clinically significant abnormality, including serum chemistry, hematology, coagulation, and urinalysis test values (abnormal tests may be repeated for confirmation)

  * Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (83):
- United States (32):
  - Teva Investigational Site 13834, Phoenix, Arizona
  - Teva Investigational Site 13819, Canoga Park, California
  - Teva Investigational Site 13811, Santa Monica, California
  - Teva Investigational Site 13823, Stanford, California
  - Teva Investigational Site 13837, Aurora, Colorado
  - Teva Investigational Site 13814, Colorado Springs, Colorado
  - Teva Investigational Site 13836, Denver, Colorado
  - Teva Investigational Site 13813, Englewood, Colorado
  - Teva Investigational Site 13821, New Haven, Connecticut
  - Teva Investigational Site 13812, Stamford, Connecticut
  - Teva Investigational Site 13810, Gainesville, Florida
  - Teva Investigational Site 13815, Orlando, Florida
  - Teva Investigational Site 13829, Ormond Beach, Florida
  - Teva Investigational Site 13830, St. Petersburg, Florida
  - Teva Investigational Site 13842, Tampa, Florida
  - Teva Investigational Site 13840, Tampa, Florida
  - Teva Investigational Site 13833, Columbus, Georgia
  - Teva Investigational Site 13826, Chicago, Illinois
  - Teva Investigational Site 13818, Ann Arbor, Michigan
  - Teva Investigational Site 13835, Las Vegas, Nevada
  - Teva Investigational Site 13832, Las Vegas, Nevada
  - Teva Investigational Site 13831, Lebanon, New Hampshire
  - Teva Investigational Site 13820, Princeton, New Jersey
  - Teva Investigational Site 13827, Albuquerque, New Mexico
  - Teva Investigational Site 13816, Amherst, New York
  - Teva Investigational Site 13817, New York, New York
  - Teva Investigational Site 13809, Raleigh, North Carolina
  - Teva Investigational Site 13839, Salisbury, North Carolina
  - Teva Investigational Site 13825, Cleveland, Ohio
  - Teva Investigational Site 13824, Philadelphia, Pennsylvania
  - Teva Investigational Site 13841, Richmond, Texas
  - Teva Investigational Site 13822, Virginia Beach, Virginia
- Australia (5):
  - Teva Investigational Site 78120, Auchenflower
  - Teva Investigational Site 78118, Clayton
  - Teva Investigational Site 78123, Melbourne
  - Teva Investigational Site 78122, Parkville
  - Teva Investigational Site 78121, Randwick
- Canada (2):
  - Teva Investigational Site 11132, Newmarket, Ontario
  - Teva Investigational Site 11130, Calgary
- Finland (3):
  - Teva Investigational Site 40030, Helsinki
  - Teva Investigational Site 40031, Oulu
  - Teva Investigational Site 40029, Turku
- Germany (7):
  - Teva Investigational Site 32666, Berlin
  - Teva Investigational Site 32667, Bochum
  - Teva Investigational Site 32660, Essen
  - Teva Investigational Site 32665, Hamburg
  - Teva Investigational Site 32662, Kiel
  - Teva Investigational Site 32661, Königstein im Taunus
  - Teva Investigational Site 32663, Rostock
- Israel (8):
  - Teva Investigational Site 80124, Ashkelon
  - Teva Investigational Site 80122, Hadera
  - Teva Investigational Site 80125, Holon
  - Teva Investigational Site 80121, Jerusalem
  - Teva Investigational Site 80123, Netanya
  - Teva Investigational Site 80120, Ramat Gan
  - Teva Investigational Site 80127, Tel Aviv
  - Teva Investigational Site 80126, Tel Aviv
- Italy (6):
  - Teva Investigational Site 30190, Milan
  - Teva Investigational Site 30192, Modena
  - Teva Investigational Site 30194, Napoli
  - Teva Investigational Site 30193, Pavia
  - Teva Investigational Site 30191, Rome
  - Teva Investigational Site 30189, Rome
- Netherlands (3):
  - Teva Investigational Site 38118, Leiden
  - Teva Investigational Site 38119, Nijmegen
  - Teva Investigational Site 38117, Zwolle
- Poland (5):
  - Teva Investigational Site 53380, Bialystok
  - Teva Investigational Site 53383, Krakow
  - Teva Investigational Site 53379, Krakow
  - Teva Investigational Site 53382, Lodz
  - Teva Investigational Site 53381, Szczecin
- Spain (5):
  - Teva Investigational Site 31211, Galdakao
  - Teva Investigational Site 31214, Madrid
  - Teva Investigational Site 31213, Seville
  - Teva Investigational Site 31212, Valladolid
  - Teva Investigational Site 31215, Zaragoza
- Sweden (2):
  - Teva Investigational Site 42047, Huddinge
  - Teva Investigational Site 42045, Vällingby
- United Kingdom (5):
  - Teva Investigational Site 34224, Glasgow
  - Teva Investigational Site 34222, Liverpool
  - Teva Investigational Site 34223, London
  - Teva Investigational Site 34220, London
  - Teva Investigational Site 34221, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 275 participants with episodic cluster headache (ECH) or chronic cluster headache (CCH) were enrolled in this study.
Pre-assignment Details: Participants were assigned to receive treatments in fremanezumab 225 milligrams (mg) monthly, fremanezumab 675/225 mg monthly, or fremanezumab 675 mg quarterly groups; based on their randomization in the pivotal studies TV48125-CNS-30056 (NCT02945046) and TV48125-CNS-30057 (NCT02964338).
Groups:
- Fremanezumab 225 mg Monthly: Participants with ECH or CCH who received fremanezumab at 900 mg intravenous (IV) infusion at Week 0 and fremanezumab at 225 mg subcutaneous (SC) injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30056 or TV48125-CNS-30057, and participants with CCH who received fremanezumab at 675 mg SC injection at Week 0 and fremanezumab at 225 mg SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30057; received fremanezumab at 225 mg SC injection monthly (approximately every 4 weeks, administered as single SC injection of fremanezumab at 225 mg [225 mg/1.5 milliliter {mL}] at Week 0 and 36; and 2 placebo SC injections at Weeks 0, 12, 24, and 36 for blinding in participants rolled over from Study TV48125-CNS-30056; fremanezumab at 225 mg as a single SC injection [225 mg/1.5 mL] at Week 0, 12, 24, and 36; 2 SC injections of placebo at Week 0 for blinding in participants rolled over from Study TV48125-CNS-30057) through Week 36 in this study.
- Fremanezumab 675/225 mg Monthly: Participants with CCH who received placebo IV infusion and SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30057; received fremanezumab 675 mg SC injection as loading dose (administered as 3 SC injections of fremanezumab at 225 mg [225 mg/1.5 mL] at Week 0) followed by monthly (approximately every 4 weeks) fremanezumab at 225 mg SC injection (administered as single SC injection of fremanezumab at 225 mg [225 mg/1.5 mL] at Weeks 12, 24, and 36) through Week 36.
- Fremanezumab 675 mg Quarterly: Participants with ECH who received fremanezumab at 675 mg SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study; or placebo IV infusion and SC injection at Week 0 and placebo SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30056; received fremanezumab at 675 mg SC injection quarterly (approximately every 12 weeks, administered as 3 SC injections of fremanezumab at 225 mg [225 mg/1.5 mL] at Weeks 0 and 36; and single placebo SC injection at Weeks 4, 8, 16, 20, 28, and 32 for blinding) through Week 36.
Period: Overall Study
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Started (Intent-to-treat (ITT) analysis set: all participants enrolled for long-term safety evaluation) | 145 | 60 | 70
Safety Analysis Set (All participants who received at least 1 dose of study drug) | 144 (1 participant assigned to 225 mg monthly arm but received 675 mg quarterly after >12 weeks remission) | 60 | 71 (1 participant assigned to 225 mg monthly arm but received 675 mg quarterly after >12 weeks remission)
Completed | 26 | 14 | 29
Not Completed | 119 | 46 | 41
Not completed — Adverse Event | 6 | 1 | 2
Not completed — Withdrawal by Subject | 9 | 5 | 8
Not completed — Protocol Violation | 6 | 0 | 3
Not completed — Lost to Follow-up | 4 | 0 | 1
Not completed — Lack of Efficacy | 23 | 7 | 4
Not completed — Other than specified | 4 | 2 | 0
Not completed — Study terminated due to futility | 67 | 31 | 23

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all participants who were enrolled in this study for long-term safety evaluation, regardless if they received study treatment or not.
Groups:
- Fremanezumab 225 mg Monthly: Participants with ECH or CCH who received fremanezumab at 900 mg IV infusion at Week 0 and fremanezumab at 225 mg SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30056 or TV48125-CNS-30057, and participants with CCH who received fremanezumab at 675 mg SC injection at Week 0 and fremanezumab at 225 mg SC injection at Weeks 4 and 8, respectively in the pivotal study TV48125-CNS-30057; received fremanezumab at 225 mg SC injection monthly (approximately every 4 weeks, administered as single SC injection of fremanezumab at 225 mg [225 mg/1.5 mL] at Week 0 and 36; and 2 placebo SC injections at Weeks 0, 12, 24, and 36 for blinding in participants rolled over from Study TV48125-CNS-30056; fremanezumab at 225 mg as a single SC injection [225 mg/1.5 mL] at Week 0, 12, 24, and 36; 2 SC injections of placebo at Week 0 for blinding in participants rolled over from Study TV48125-CNS-30057) through Week 36 in this study.
- Total: Total of all reporting groups
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly | Total
Number analyzed (Participants) | 145 | 60 | 70 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.25) | 46.1 (11.14) | 43.2 (11.40) | 44.9 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 20 | 25 | 96
  Male | 94 | 40 | 45 | 179
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 3 | 2 | 14
  White | 136 | 56 | 68 | 260
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to follow-up (Week 68)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 144 | 60 | 71
Participants
  Any AEs | 87 | 31 | 42
  Treatment-related AEs | 26 | 6 | 10
  Serious AEs | 8 | 2 | 1
  AEs leading to discontinuation | 6 | 1 | 2

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Results: Serum Chemistry
Description: Serum chemistry tests with potentially clinically significant abnormal findings included: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), lactate dehydrogenase (LDH) each ≥3*upper limit of normal (ULN); Blood urea nitrogen (BUN) ≥10.71 millimole (mmol)/L; Bilirubin (Total) ≥34.2 micromole/liter (umol/L); and Creatinine ≥177 umol/L. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to end of treatment (Week 40)
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants with a laboratory result.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 129 | 55 | 67
Participants | 2 | 0 | 1

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Results: Hematology
Description: Hematology tests with potentially clinically significant abnormal findings included: hemoglobin less than or equal to (≤)115 grams (g)/L (males) or ≤95 g/L (females), leukocytes count ≥20*10^9/L or ≤3*10^9/L, eosinophils ≥10%, hematocrit <0.37 L/L (males) and <0.32 L/L (females), platelets count ≥700*10^9/L or ≤75*10^9/L, absolute neutrophil count (ANC) ≤1*10^9/L. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to end of treatment (Week 40)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 129 | 55 | 67
Participants | 6 | 3 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Results: Urinalysis
Description: Urinalysis laboratory tests with potentially clinically significant abnormal findings included: haemoglobin, urine glucose, ketones, urine total protein each ≥2 unit (U) increase from baseline. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to end of treatment (Week 40)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 129 | 55 | 67
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Shift From Baseline to Endpoint (Last Assessment) in Coagulation Laboratory Test Results
Description: Coagulation parameters included: prothrombin time (PT) (seconds) and prothrombin international normalized ratio (INR). Shifts represented as Baseline - endpoint value (last observed post-baseline value). Shifts from baseline to endpoint were summarized using participant counts grouped into three categories: - Low (below normal range) - Normal (within the normal range of 9.4 to 12.5 seconds) - High (above normal range). Missing PT and prothrombin INR shift data are also presented. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to end of treatment (Week 40)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 144 | 60 | 71
Participants
  Prothrombin INR: Low-Low | 0 | 0 | 0
  Prothrombin INR: Low-Normal | 0 | 0 | 0
  Prothrombin INR: Low-High | 0 | 0 | 0
  Prothrombin INR: Normal-Low | 1 | 0 | 0
  Prothrombin INR: Normal-Normal | 103 | 42 | 61
  Prothrombin INR: Normal-High | 6 | 4 | 1
  Prothrombin INR: High-Low | 0 | 0 | 0
  Prothrombin INR: High-Normal | 7 | 4 | 3
  Prothrombin INR: High-High | 4 | 2 | 0
  Prothrombin INR: Missing | 23 | 8 | 6
  PT: Low-Low | 0 | 0 | 0
  PT: Low-Normal | 0 | 0 | 0
  PT: Low-High | 0 | 0 | 0
  PT: Normal-Low | 1 | 0 | 0
  PT: Normal-Normal | 99 | 39 | 59
  PT: Normal-High | 6 | 5 | 1
  PT: High-Low | 0 | 0 | 0
  PT: High-Normal | 11 | 4 | 5
  PT: High-High | 4 | 4 | 0
  PT: Missing | 23 | 8 | 6

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Potentially clinically significant abnormal vital signs findings included: Pulse rate ≥120 beats per minute (bpm) and increase from baseline of ≥15 bpm, or ≤50 bpm and decrease from baseline of ≥15 bpm; Systolic blood pressure ≤90 millimeters of mercury (mmHg) and decrease from baseline of ≥20 mmHg, or ≥180 mmHg and increase from baseline of ≥20 mmHg; Diastolic blood pressure ≤50 mmHg and decrease from baseline of ≥15 mmHg, or ≥105 mmHg and increase from baseline of ≥15 mmHg; Temperature >38.3 degrees celsius (°C). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to follow-up (Week 68)
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants with a vital sign result.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 139 | 57 | 68
Participants | 6 | 4 | 2

7. Primary Outcome: Number of Participants With Shift From Baseline to Endpoint (Last Assessment) in Electrocardiogram (ECG) Parameters
Description: ECG parameters included: heart rate, PR interval, QRS interval, QT interval corrected using the Fridericia formula (QTcF), QT interval corrected using the Bazett's formula (QTcB) and RR interval. Shifts represented as Baseline - endpoint value (last observed post-baseline value). Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding. Missing ECG shift data are also presented. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to follow-up (Week 68)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 144 | 60 | 71
Participants
  Normal / Normal | 76 | 30 | 46
  Normal / Abnormal NCS | 16 | 6 | 4
  Normal / Abnormal CS | 1 | 0 | 0
  Abnormal NCS / Normal | 15 | 7 | 4
  Abnormal NCS / Abnormal NCS | 23 | 12 | 12
  Abnormal NCS / Abnormal CS | 0 | 0 | 0
  Abnormal CS / Normal | 0 | 0 | 0
  Abnormal CS / Abnormal NCS | 0 | 0 | 0
  Abnormal CS / Abnormal CS | 0 | 0 | 0
  Missing | 13 | 5 | 5

8. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: A complete physical examination included the following organ systems: general appearance; head, eyes, ears, nose, and throat; chest and lungs; heart; abdomen; musculoskeletal; skin; lymph nodes; and neurological. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to follow-up (Week 68)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 145 | 60 | 70
Participants | 22 | 8 | 7

9. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Number of participants who reported treatment-emergent injection site reactions are summarized. Preferred terms from Medical Dictionary for Regulatory Activities (MedDRA) version 18.1 were offered without a threshold applied. Injection site reactions included injection site erythema, induration, pain, haemorrhage, bruising, rash, warmth, and pruritus. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to Week 36
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 144 | 60 | 71
Participants
  Injection site induration | 13 | 4 | 5
  Injection site pain | 6 | 1 | 3
  Injection site erythema | 7 | 1 | 1
  Injection site haemorrhage | 2 | 0 | 0
  Injection site pruritus | 2 | 0 | 0
  Injection site bruising | 0 | 1 | 0
  Injection site rash | 0 | 0 | 1
  Injection site warmth | 1 | 0 | 0

10. Primary Outcome: Number of Participants With Hypersensitivity/Anaphylaxis Reactions
Description: A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to Week 36
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 144 | 60 | 71
Participants | 0 | 0 | 0

11. Primary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medications included: agents acting on the renin-angiotensin system, all other therapeutic products (homeopathic), allergens, analgesics, anesthetics, anti-parkinson drugs, antianemic preparations, antibacterials, antibiotics and chemotherapeutics for dermatological use, antidiarrheals, intestinal antiinflammatory/antiinfective agents, antiemetic, antiepileptics, antifungals for dermatologiocal use, antigout preparations, antihemorrhagics, antihistamines for systemic use, antihypertensives, antiinflammatory and antirheumatic products, antimycotics for systemic use, antipruritics, antipsoriatics, antivirals for systemic use, beta blocking agents, blood substitutes and perfusion solutions, cardiac therapy, corticosteroids, cough and cold preparations, diagnostic radiopharmaceuticals, diuretics, thyroid therapy, urologicals, vaccines, psycoleptics, psycoanaleptics, ophthalmologicals, muscle relaxants, drugs used in diabetes. Baseline refers to values from the pivotal studies.
Time Frame: Baseline up to follow-up (Week 68)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 144 | 60 | 71
Participants | 140 | 56 | 68

12. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior as Assessed by the Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
Description: eC-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent. Baseline refers to the baseline values from the pivotal studies.
Time Frame: Baseline up to follow-up (Week 68)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
Number analyzed (Participants) | 145 | 60 | 70
Participants | 7 | 1 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 68
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | Fremanezumab 225 mg Monthly | Fremanezumab 675/225 mg Monthly | Fremanezumab 675 mg Quarterly
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/60 | 0/71
Serious Adverse Events (participants affected / at risk) | 8/144 | 2/60 | 1/71
Other Adverse Events (participants affected / at risk) | 31/144 | 11/60 | 14/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fremanezumab 225 mg Monthly (N=144) | Fremanezumab 675/225 mg Monthly (N=60) | Fremanezumab 675 mg Quarterly (N=71)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fremanezumab 225 mg Monthly (N=144) | Fremanezumab 675/225 mg Monthly (N=60) | Fremanezumab 675 mg Quarterly (N=71)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 0 (0)
Injection site induration (General disorders) | 13 (44) | 4 (13) | 5 (10)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 16 (18) | 5 (8) | 7 (8)
Sinusitis (Infections and infestations) | 4 (4) | 3 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated after the ECH study (TV48125-CNS-30056) was terminated due to a pre specified futility analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT03107052/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT03107052/SAP_001.pdf